CLINICAL TRIAL: NCT04842630
Title: An Open-Label, Multicenter, Dose Escalation And Expansion Study Of SHR-1916 In Subjects With Locally Advanced Or Metastatic Solid Tumor Malignancies
Brief Title: A Phase 1 Dose Escalation and Expansion Study Of SHR-1916 In Subjects With Locally Advanced Or Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: R&d strategy adjustment
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1916-I-101
Record Dates: First submitted 2021-04-01; First posted 2021-04-13 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1916 (Experimental)
  Interventions: Drug: SHR-1916

INTERVENTIONS:
Drug: SHR-1916 — All participants receive SHR-1906 alone

SUMMARY:
This is a first in human, open-label, dose escalation and expansion Phase 1 study of SHR-1916 in adult patients with locally advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and the willingness to sign a written informed consent document；
2. Aged between 18-75 years old;
3. Histologically or cytologically confirmed advanced or metastatic malignant tumor;
4. Presence of at least of one measurable lesion in agreement to RECIST criteria;
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1;
6. Life expectancy >12 weeks;
7. Adequate organ performance based on laboratory blood tests;
8. Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation.

Exclusion Criteria:

1. Patients who have received cytokines (IL-2, IFN-α)as anti-tumor therapy within 6 months before the first dose;
2. Previous systemic therapy within 28 days before the first dose;
3. Previous therapeutic surgery within 28 days, and diagnostic surgery within 14 days prior to the first dose;
4. Received live attenuated vaccine within 28 days before the first dose, or expected to receive live attenuated vaccine during the study treatment period;
5. Patients who received systemic immunosuppressive therapy within 14 days before the first dose;
6. Patients with known or suspected brain metastasis；
7. Subjects with interstitial pneumonia or interstitial lung disease, with a history of interstitial pneumonia or interstitial lung disease limiting self care ADL or with life-threatening respiratory compromise, with a history of pulmonary fibrosis, lasting pneumonia, drug- or radiation-induced pneumonia, and congenital pneumonia that may otherwise interfere with the judgement of immune-related pulmonary toxicity, or with any evidence of active pneumonia as shown on chest CT scans;
8. Patients with history of autoimmune diseases;
9. History of immunodeficiency (including HIV infection) or organ transplantation;
10. Known active hepatitis B or C infection;
11. Other serious accompanying illnesses, which, in the researcher's opinion, could seriously adversely affect the safety of the treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Dose Limited Toxicity (DLT) | 21 Days (first cycle)
Maximum tolerable dose (MTD) | 21 Days (first cycle)
Recommended dose for phase II (RP2D) | Up to 8 months

SECONDARY OUTCOMES:
AEs （Adverse Events） | 30 days after last dose
Area under the plasma concentration time curve in the dosing interval AUC(TAU) of SHR-1916 | 30 days after last dose
Maximum observed plasma concentration (Cmax) of SHR-1916 | 30 days after last dose
Minimum observed plasma concentration (Cmin) of SHR-1916 | 30 days after last dose
Time of maximum observed plasma concentration (Tmax) of SHR-1916 | 30 days after last dose
Percentage of NK cell and CD8+ T cell by flow cytometry | 30 days after last dose
Absolute count values of NK cell and CD8+ T cell by flow cytometry | 30 days after last dose
Peripheral plasma concentration of sCD25 | 30 days after last dose
Immunogenicity analysis to assess anti-drug antibodies (ADA) to SHR-1916 in human serum | 30 days after last dose
ORR（Objective Response Rate） | at the time point of every 9 weeks
DCR（Disease Control Rate） | at the time point of every 9 weeks
DoR（Duration of Response） | up to 2 years
PFS（Progression-Free-Survival） | up to 2 years
12-month-survival Rate | up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China